CLINICAL TRIAL: NCT01979757
Title: Outcomes After Centrifugation Versus PureGraft for Fatgrafting to the Breast After Breast-conserving Therapy
Brief Title: Outcomes After Centrifugation Versus PureGraft for Fatgrafting to the Breast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulovka Hospital (Other)
Responsible Party: Principal Investigator, Ondrej Mestak M.D., Consultant, Bulovka Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CentPure; 268011 (Other Grant/Funding Number: Grant Agency of Charles University in Prague)
Record Dates: First submitted 2013-10-28; First posted 2013-11-08 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Fatgrafting to a Breast After Breast Conserving Therapy
MeSH Terms: interventions — Centrifugation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Centrifugation (Active Comparator): Patients recieved fatgraft processed by Centrifugation
  Interventions: Other: Centrifugation
- Puregraft (Active Comparator): Patients recieved fatgraft processed by Puregraft
  Interventions: Other: Puregraft

INTERVENTIONS:
Other: Puregraft
  Arms: Puregraft
Other: Centrifugation
  Arms: Centrifugation

SUMMARY:
Breast-conserving treatment (BCT) leads to a progressive and deteriorating breast deformity. Fatgrafting is ideal for breast reconstruction after BCT. The most frequently utilized technique for fat processing is centrifugation. The PureGraft device (Cytori Therapeutics, USA) is a new method that involves washing and filtering the fat to prepare the graft. The investigators compared the subjective and objective outcomes of two fat-processing methods, centrifugation and PureGraft filtration.

Thirty patients underwent breast reconstruction performed by a single surgeon (OM) after BCT in our department between April 2011 and September 2012. The patients were preoperatively divided into two groups randomly: 15 received fatgrafts processed by centrifugation, and 15 received fatgrafts processed by washing in PureGraft bags. The patients were followed up for 12-30 months.To measure the subjective outcome, the investigators distributed the BREAST-Q questionnaire to all the patients both preoperatively and one year postoperatively. The BCCT.core software evaluated the objective outcome of breast reconstruction by fatgrafting.

ELIGIBILITY:
Inclusion Criteria:

* State after breast conserving therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Outcomes after centrifugation versus PureGraft for fatgrafting to the breast after breast-conserving therapy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ondrej Mestak, M.D., Study Chair — Charles University, Czech Republic
Locations (1):
- Bulovka Hospital, Prague, Czechia